CLINICAL TRIAL: NCT02559687
Title: A Phase II Study of Pembrolizumab Monotherapy in Third Line Previously Treated Subjects With Advanced/Metastatic Adenocarcinoma or Squamous Cell Carcinoma of the Esophagus or Advanced/Metastatic Siewert Type I Adenocarcinoma of the Esophagogastric Junction (KEYNOTE-180)
Brief Title: Study of Pembrolizumab (MK-3475) in Previously-Treated Participants With Advanced Carcinoma of the Esophagus or Esophagogastric Junction (MK-3475-180/KEYNOTE-180)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-180; 163188 (Registry Identifier: JAPIC-CTI); MK-3475-180 (Other: Merck); KEYNOTE -180 (Other: Merck); 2015-002427-26 (EudraCT Number)
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Carcinoma; Esophagogastric Junction Carcinoma
Keywords: Programmed Cell Death-1 (PD-1, PD1); Programmed Cell Death-Ligand 1 (PD-L1, PDL1); Programmed Cell Death-Ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Esophageal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pembrolizumab 200 mg (Experimental): Participants will receive pembrolizumab 200 mg, intravenously (IV), every 3 weeks (Q3W) for up to 35 treatments (approximately 2 years). Eligible participants who stop pembrolizumab with Stable Disease (SD) or better but progress after discontinuation may be able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
  Interventions: Biological: pembrolizumab

INTERVENTIONS:
Biological: pembrolizumab — IV Q3W
  Other Names: MK-3475

SUMMARY:
In this study participants with advanced/metastatic adenocarcinoma of the esophagus (EAC), squamous cell carcinoma of the esophagus (ESCC), or advanced/metastatic Siewert type I adenocarcinoma of the esophagogastric junction (EGJ), who had been previously treated with two standard therapies, will be treated with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than 3 months
* Histologically-proven advanced/metastatic adenocarcinoma or squamous cell carcinoma of the esophagus or advanced/metastatic Siewert type 1 adenocarcinoma of the EGJ
* Documented objective radiographic or clinical disease progression on two previous lines of standard therapy
* Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* Can provide either a newly obtained or archival tumor tissue sample for intratumoral immune-related testing and for anti-programmed cell death (PD-1)
* Female participants of childbearing potential must be willing to use adequate contraception for the course of the study through 120 days after the last dose of study medication
* Male participants must agree to use adequate contraception starting with the first dose through 120 days after the last dose of study medication
* Adequate organ function

Exclusion Criteria:

* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study medication
* Has active autoimmune disease that has required systemic treatment within the 2 years prior to the first dose of study medication
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Prior anti-cancer mAb, chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to first dose of study medication or not recovered from adverse events due to a previously administered agent
* Prior therapy with an anti-PD-1, anti-PD-Ligand 1 (PD-L1), or anti-PD-L2 agent, or previously participated in a Merck pembrolizumab (MK-3475) study
* Has a known additional malignancy that has progressed or required active treatment within the last 5 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, in-situ cervical cancer, and in-situ or intra-mucosal pharyngeal cancer
* Received a live vaccine within 30 days of the first dose of study medication
* Known history of Human Immunodeficiency Virus (HIV) infection
* Known active Hepatitis B or C
* History of non-infectious pneumonitis that required steroids or current pneumonitis
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Shah MA, Kojima T, Hochhauser D, Enzinger P, Raimbourg J, Hollebecque A, Lordick F, Kim SB, Tajika M, Lockhart AC, Arkenau HT, El-Hajbi F, Gupta M, Pfeiffer P, Bhagia P, Cao ZA, Lunceford J, Suryawanshi S, Ayers M, J Marton M, Kato K. T cell-inflamed gene expression profile and PD-L1 expression and pembrolizumab efficacy in advanced esophageal cancer. Future Oncol. 2022 Jul 19. doi: 10.2217/fon-2021-1134. Online ahead of print. PMID 35852104
- [Derived] Shah MA, Kojima T, Hochhauser D, Enzinger P, Raimbourg J, Hollebecque A, Lordick F, Kim SB, Tajika M, Kim HT, Lockhart AC, Arkenau HT, El-Hajbi F, Gupta M, Pfeiffer P, Liu Q, Lunceford J, Kang SP, Bhagia P, Kato K. Efficacy and Safety of Pembrolizumab for Heavily Pretreated Patients With Advanced, Metastatic Adenocarcinoma or Squamous Cell Carcinoma of the Esophagus: The Phase 2 KEYNOTE-180 Study. JAMA Oncol. 2019 Apr 1;5(4):546-550. doi: 10.1001/jamaoncol.2018.5441. PMID 30570649
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 185 participants screened for inclusion, 121 were enrolled and received treatment. Per protocol, response/progression or adverse events (AEs) that occurred during the second course were not counted towards efficacy outcome measures or safety outcome measures, respectively.
Groups:
- Pembrolizumab 200 mg: Participants received pembrolizumab 200 mg, intravenously (IV), every 3 weeks (Q3W) for up to 35 treatments (approximately 2 years). Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
Period: Overall Study
Arm/Group | Pembrolizumab 200 mg
Started | 121
Received First Course of Pembrolizumab | 121
Received Second Course of Pembrolizumab | 1
Completed | 0
Not Completed | 121
Not completed — Death | 112
Not completed — Sponsor Decision | 5
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 42
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 71
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) According to Response Evaluation Criteria for Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experienced a CR or PR based on modified RECIST 1.1 was reported per protocol for the first course of treatment.
Time Frame: Up to approximately 28 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pembrolizumab 200 mg: Participants receive pembrolizumab 200 mg IV Q3W for up to 35 treatments (approximately 2 years).
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 121
percentage of participants | 9.9 [5.2 to 16.7]

2. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product, was also an adverse event. The number of participants who experienced ≥1 AE was reported per protocol for the first course of treatment.
Time Frame: Up to approximately 59 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 121
Participants | 116

3. Secondary Outcome: Number of Participants That Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product, was also an adverse event. The number of participants that discontinued study treatment due to an AE was reported per protocol for the first course of treatment.
Time Frame: Up to approximately 24 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 121
Participants | 14

4. Secondary Outcome: Duration of Response (DOR) According to RECIST 1.1 Assessed by BICR
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. DOR assessments were based on blinded central imaging review with confirmation. The DOR per RECIST 1.1 for all participants who experienced a confirmed CR or PR was reported per protocol for the first course of treatment.
Time Frame: Up to approximately 67 months
Population: All allocated participants who received at least 1 dose of study treatment and who experienced a confirmed CR or confirmed PR. One previously reported participant was excluded from the DOR analysis based on a BICR re-read of prior scans after the primary analysis database lock.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 11
Months | 19.7 [2.1 to 60.3]

5. Secondary Outcome: Progression Free Survival (PFS) According to RECIST 1.1 Assessed by BICR
Description: PFS was defined as the time from first day of study treatment to the first documented PD or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of ≥1 new lesions was also considered PD. PFS as assessed by blinded independent central review per RECIST 1.1 was reported per protocol for the first course of treatment.
Time Frame: Up to approximately 67 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 121
Months | 2.0 [1.9 to 2.1]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first day of study treatment to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS was reported per protocol for the first course of treatment
Time Frame: Up to approximately 67 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 121
Months | 5.8 [4.5 to 7.2]

ADVERSE EVENTS:
Time Frame: Up to approximately 67 months
Description: All-Cause Mortality was reported for all allocated participants.
  Serious AEs and Other AEs were reported for all allocated participants who received at least 1 dose of study treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Pembrolizumab 200 mg First Course: Participants received pembrolizumab 200 mg IV Q3W for up to 35 treatments (approximately 2 years).
- Pembrolizumab 200 mg Second Course: Eligible participants who stopped the initial course of pembrolizumab (200 mg IV Q3W for up to 35 treatments [approximately 2 years]) with Stable Disease (SD) or better but progressed after discontinuation initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (up to approximately 1 additional year).
Arm/Group | Pembrolizumab 200 mg First Course | Pembrolizumab 200 mg Second Course
All-Cause Mortality (participants affected / at risk) | 116/121 | 0/1
Serious Adverse Events (participants affected / at risk) | 47/121 | 0/1
Other Adverse Events (participants affected / at risk) | 107/121 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg First Course (N=121) | Pembrolizumab 200 mg Second Course (N=1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 2 (2) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 16 (17) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 5 (5) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg First Course (N=121) | Pembrolizumab 200 mg Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 18 (22) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 11 (13) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 0 (0)
Constipation (Gastrointestinal disorders) | 23 (24) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 18 (22) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 8 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 22 (26) | 0 (0)
Oral pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 19 (25) | 0 (0)
Asthenia (General disorders) | 9 (10) | 0 (0)
Fatigue (General disorders) | 34 (37) | 0 (0)
Oedema peripheral (General disorders) | 10 (11) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 8 (13) | 1 (1)
Pneumonia (Infections and infestations) | 9 (9) | 0 (0)
Alanine aminotransferase increased (Investigations) | 12 (13) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 13 (14) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 10 (11) | 0 (0)
Blood bilirubin increased (Investigations) | 9 (9) | 0 (0)
Weight decreased (Investigations) | 7 (8) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 23 (23) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (10) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (8) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (13) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 7 (7) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (10) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (13) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 10 (13) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT02559687/Prot_SAP_001.pdf